CLINICAL TRIAL: NCT05560074
Title: The Effect of Two Different Non-pharmacologic Methods (Buzzy® and DistrACTION® Cards) for Pain and Fear Relief During Blood Specimen Collection in Children: A Randomized Controlled Trial
Brief Title: The Effect of Two Different Non-pharmacologic Methods for Painandfear Relief During Blood Specimen Collection Inchildren
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Tübingen University
Record Dates: First submitted 2022-08-22; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-08

CONDITIONS: Pain
Keywords: Pain; children; buzzy; distractionCards; blood sample
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Buzzy (Experimental): Buzzy®: It is a 8x5x2.5 cm sized, noninvasive device used for pain control in adults and children, developed by the pediatrician Ammy Baxter, with a plastic battery and vibration motor. A cold ice pack is placed under Buzzy. It has a local cold application and vibration effect. It is placed 3~5 cm above the injection site for 15~30 sec before and during the procedure, making local cold application and vibrations. One should be sure about the definite contact of Buzzy® with the skin. The ice pack is kept in a deep freezer and placed in the device before the procedure. After the procedure is completed, the ice pack is wiped with 70% alcohol, and kept and chilled again in the deep freezer. http://www.buzzy4shots.com/)
  Interventions: Device: Buzzy
- DistractionCards (Experimental): DistrACTION® Cards consisted of visual cards of 5 cm × 8 cm, covered with various pictures and shapes. In this method, the children first carefully examine the cards. Then, the PhD-qualified nurse researcher asks some questions about those cards to be answered by the children, such as "How many ladybugs are there in the picture?" "How many apes are there in the picture?" or "Can you see the comet?" The distraction procedure via distraction cards begin just before the venous blood specimen collection and continue until the end of the blood specimen collection
  Interventions: Other: DistrACTION® Cards
- Control (No Intervention): Controll group: Venous blood will be taken as usual on the blood collection room without applying an intervention to the children in the Control group. Children will follow the standard blood draw procedure.

INTERVENTIONS:
Device: Buzzy — In the Buzzy® group, 30 seconds before the blood collection procedure and during the procedure, the Buzzy® device ist placed 3-5 cm above the area from where the blood would be taken by the PhD qualified nurse researcher
  Arms: Buzzy
Other: DistrACTION® Cards — In the DistrACTION® Cards group, picture cards containing various hidden pictures and patterns are used during blood collection by the PhD qualified nurse researcher
  Arms: DistractionCards

SUMMARY:
Introduction: Pain is defined as an unpleasant emotional and sensorial feeling that arises from any part of the body progresses with possible tissue damage and covers all past experiences of individuals.

The aim of this randomized-controlled study is to compare the effect of two methods (Buzzy® and DistrACTION® Cards) used to reduce pain and anxiety during blood specimen collection in children.

Material and Methods: Children between the ages of 6 and 12 who come to the Tübingen University Rheumatology outpatient clinic will be included in the study.

Keywords: Pain, children, blood sample Research Hypotheses Hypothesis 0 (H0):There is no difference in terms of procedural pain and anxiety between children in the control group and interventions groups (Buzzy®, DistraCTION® Cards).

Hypothesis 1 (H1): Children who received Buzzy® during venous blood specimen collection have less pain and anxiety than children in the control group.

Hypothesis 2 (H2): Children who received DistrACTION® Cards during venous blood specimen collection have less pain and anxiety than children in the control group.

Hypothesis 3 (H3): Children who received Buzzy® during venous blood specimen collection have less pain and anxiety than children in the DistrACTION® Cards group.

In the study, we will use an information form that involves questions about the descriptive characteristics of the children and their families (parents' educational level, age, gender) and the blood specimen collection process (past and present experience), child's body mass index (BMI), the Children's Fear Scale (CFS) to determine the anxiety of the children and Faces Pain Scale-Revised (FPS-R) to evaluate pain. A pilot will be used to test whether the questions are understood before the questionnaires are administered.

Keywords: Pain, children, blood sample, buzzy, distractionCards

DETAILED DESCRIPTION:
The study will be carried out with the children and their parents who come to the rheumatology outpatient clinic at the University Hospital Tuebingen with their parents and met the sampling selection criteria.

An information letter describing the research study will be sent to the addresses of children and their families who meet the criteria before they come to the outpatient department.

When the child and parent come to the outpatient appointment:

* The study will begin after a doctor's examination, whose blood is decided to be drawn. Blood collection will be done in a separate room.
* The researcher will explain the study herself to the child (6-12 years old) and parents. First of all, the parents and children will be informed about the research via the "Information and Consent Form" (Appendix-2,3,4,5) and will be included in the study if they wish to participate. All participants will be informed about the possibility to withdraw their participation. Only participants who have received written and verbal consent to participate in the study will be included.
* According to the computer program (from 1 to 99), blood collection from the children will be done by the researcher herself, according to the order determined by the randomization.

Course of the study control and intervention group and examination methods:

1. All groups:

   Before the venous blood collection: The parents and their children are informed about the procedures and their written and verbal consent are received. Randomization is performed. Socio-demographic information form is filled in. The children, parents, and researcher are asked to evaluate the child's level of fear using the CFS.
2. Intervention and Control:

During the venous blood collection: The blood collection procedure of all children participating in the study is performed by a PhD qualified nurse researcher experienced in blood collection using a 21-G vacuum blood collection tube needle tip from the arm. To avoid bias which can affect pain sensation or fear of the child a standardized procedure is performed during the study so that environmental bias can be excluded. The blood of the children in all groups will be taken by the same PhD qualified nurse researcher herself in the blood collection room. She will approach the children and parents in the same way and take care that the childrens perception of pain and fear is not affected by external factors.

Controll group: Venous blood will be taken as usual on the blood collection room without applying an intervention to the children in the Control group. Children will follow the standard blood draw procedure.

Intervention group 1: In the DistrACTION® Cards group, picture cards containing various hidden pictures and patterns are used during blood collection by the PhD qualified nurse researcher.

Intervention group 2: In the Buzzy® group, 30 seconds before the blood collection procedure and during the procedure, the Buzzy® device ist placed 3-5 cm above the area from where the blood would be taken by the PhD qualified nurse researcher

Data Collection Tools:

* Information form containing socio-demographics and further characteristics of the child and his family and questions on previous and current experience of the blood drawing process
* Child's pain " Faces Pain Scale-Revised (FPS-R)"
* Child's fear "Children's Fear Scale" and
* "Application Registration Form" to save the measurements made after the procedure Information form; It consists of six open and closed-ended questions about the introductory characteristics of the child and his family (parents' education level, age, gender), the blood specimen collection process (past experience), and the blood child's body mass index (BMI). In this study, the form will be filled before the blood specimen collection.

Faces Pain Scale-Revised (FPS-R) consists of six facial expressions rated from 0 to 10 according to the presence and level of pain. This scale is based on a valid and reliable personal expression in children during painful situations. In school-aged children (aged 4~12 years), the FPS-R is felt to be the most valid and reliable measure of acute pain because an understanding of words or numeric values is not needed. In the study, FPS-R are used to evaluate the children's pain after the procedure (by the children, parents, researcher).

The Children's Fear Scale (CFS) was adapted from the Faces Anxiety Scale to measure fear in children undergoing painful medical procedures. Fear facial expressions are seen from 0 to 4. These faces are showing different amounts of being scared. This face [the left-most face] is not scared at all, this face is a little bit more scared [second face from left], a bit more scared [sweep finger along scale], right up to the most scared possible [the last face on the right]. In the study, CFS are used to evaluate the children's fear before and after the procedure (by the children, parents, researcher).

ELIGIBILITY:
Inclusion Criteria:

- Children between the ages of 6-12 coming to the rheumatology outpatient clinic

Exclusion Criteria:

* having a disease that causes chronic pain,
* having a mental or neurologic disability,
* have received analgesics within the last 6 hours,
* history of fainting during blood collection,
* with cold urticaria

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Child's fear | Before and immediately after blood draw at 3-4 months
  Befor and immediately after blood draw will be assessed with Children's Fear Scale (CFS) (parent)
  The Children's Fear Scale (CFS) was adapted from the Faces Anxiety Scale to measure fear in children undergoing painful medical procedures. Fear facial expressions are seen from 0 to 4. These faces are showing different amounts of being scared. This face [the left-most face] is not scared at all, this face is a little bit more scared [second face from left], a bit more scared [sweep finger along scale], right up to the most scared possible [the last face on the right].
Change in the Child's fear | Before and immediately after blood draw at 3-4 months
  Befor and immediately after blood draw will be assessed with Children's Fear Scale (CFS) (child)
  The Children's Fear Scale (CFS) was adapted from the Faces Anxiety Scale to measure fear in children undergoing painful medical procedures. Fear facial expressions are seen from 0 to 4. These faces are showing different amounts of being scared. This face [the left-most face] is not scared at all, this face is a little bit more scared [second face from left], a bit more scared [sweep finger along scale], right up to the most scared possible [the last face on the right].
Change in the Child's fear | Before and immediately after blood draw at 3-4 months
  Befor and immediately after blood draw will be assessed with Children's Fear Scale (CFS) (researcher)
  The Children's Fear Scale (CFS) was adapted from the Faces Anxiety Scale to measure fear in children undergoing painful medical procedures. Fear facial expressions are seen from 0 to 4. These faces are showing different amounts of being scared. This face [the left-most face] is not scared at all, this face is a little bit more scared [second face from left], a bit more scared [sweep finger along scale], right up to the most scared possible [the last face on the right].

SECONDARY OUTCOMES:
Child's pain | immediately after blood draw at 3-4 months
  After blood draw will be assessed with Faces Pain Scale-Revised (FPS-R) (parent)
  Faces Pain Scale-Revised (FPS-R) consists of six facial expressions rated from 0 to 10 according to the presence and level of pain.This face [the left-most face] is not pain at all, right up to the most pain possible [the last face on the right].
Child's pain | immediately after blood draw at 3-4 months
  After blood draw will be assessed with Faces Pain Scale-Revised (FPS-R) (child)
  Faces Pain Scale-Revised (FPS-R) consists of six facial expressions rated from 0 to 10 according to the presence and level of pain.This face [the left-most face] is not pain at all, right up to the most pain possible [the last face on the right].
Child's pain | immediately after blood draw at 3-4 months
  After blood draw will be assessed with Faces Pain Scale-Revised (FPS-R)(researcher)
  Faces Pain Scale-Revised (FPS-R) consists of six facial expressions rated from 0 to 10 according to the presence and level of pain.This face [the left-most face] is not pain at all, right up to the most pain possible [the last face on the right].

CONTACTS AND LOCATIONS:
Overall Officials: Birsen Bilgen Sivri, Principal Investigator — University of Tübingen Nursing Science
Locations (1):
- University of Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
The individual information of the participants (name, surname, address,..) will not be shared. A number will be given for each.

REFERENCES:
- [Result] Sivri Bilgen B, Balci S. The Effect on Pain of Buzzy(R) and ShotBlocker(R) during the Administration of Intramuscular Injections to Children: A Randomized Controlled Trial. J Korean Acad Nurs. 2019 Aug;49(4):486-494. doi: 10.4040/jkan.2019.49.4.486. PMID 31477677
- [Result] Gerceker GO, Binay S, Bilsin E, Kahraman A, Yilmaz HB. Effects of Virtual Reality and External Cold and Vibration on Pain in 7- to 12-Year-Old Children During Phlebotomy: A Randomized Controlled Trial. J Perianesth Nurs. 2018 Dec;33(6):981-989. doi: 10.1016/j.jopan.2017.12.010. Epub 2018 Mar 17. PMID 29559294
- [Result] Ballard A, Khadra C, Adler S, Trottier ED, Le May S. Efficacy of the Buzzy Device for Pain Management During Needle-related Procedures: A Systematic Review and Meta-Analysis. Clin J Pain. 2019 Jun;35(6):532-543. doi: 10.1097/AJP.0000000000000690. PMID 30829735
- [Result] Walco GA. Needle pain in children: contextual factors. Pediatrics. 2008 Nov;122 Suppl 3:S125-9. doi: 10.1542/peds.2008-1055d. PMID 18978005
- [Result] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Result] Birnie KA, Chambers CT, Fernandez CV, Forgeron PA, Latimer MA, McGrath PJ, Cummings EA, Finley GA. Hospitalized children continue to report undertreated and preventable pain. Pain Res Manag. 2014 Jul-Aug;19(4):198-204. doi: 10.1155/2014/614784. Epub 2014 May 7. PMID 24809068
- [Derived] Bilgen Sivri B, Feng YS, Michler C, Kuemmerle-Deschner J, Mahler C. The effect of buzzy(R), DistrACTION(R) cards on reducing pediatric pain and fear during blood collection in the rheumatology polyclinic: A randomized controlled trial. J Pediatr Nurs. 2023 Nov-Dec;73:e446-e454. doi: 10.1016/j.pedn.2023.10.013. Epub 2023 Oct 31. PMID 37919179
- See also: Buzzy — http://www.buzzy4shots.com/
- See also: International Association for the Study of Pain (IASP). Pain terminology. — http://www.iasp-pain.org/Education/Content.aspx?ItemNumber=1698.